CLINICAL TRIAL: NCT04258722
Title: Reducing Adverse Delivery Outcomes Through Teleneonatology: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Samuel Gentle, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-300004483
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Newborn Morbidity
Keywords: telemedicine; simulation; neonatal resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trainee + Teleneonatologist (Experimental): Trainee, teleneonatologist, nurse, and respiratory therapist will perform resuscitation
  Interventions: Other: Resuscitation Personnel
- Trainee (Active Comparator): Trainee, nurse, and respiratory therapist will perform resuscitation.
  Interventions: Other: Resuscitation Personnel

INTERVENTIONS:
Other: Resuscitation Personnel — Type of resuscitation team

SUMMARY:
Teleneonatology, the use of audio-video communication to facilitate neonatal-perinatal care, may bridge the resuscitation quality gap by connecting centers with lower level care to experienced care providers. Using randomized trial design, this investigation will compare teleneonatal resuscitation facilitated by a neonatologist to standard resuscitation within a simulated environment.

DETAILED DESCRIPTION:
Multiple studies have evaluated telemedicine using simulation, but the level of evidence for the use of telemedicine to improve neonatal resuscitation is low.

In this investigation and within a simulated environment, pediatric interns and residents will resuscitate a simulated 25 week infant at delivery assisted by a simulated nurse and respiratory therapist. Participants will be randomized to resuscitation performed either with or without telemedicine facilitated by a neonatologist. The primary outcome will be time to effective ventilation with other secondary outcomes including metrics derived from the American Academy of Pediatrics Neonatal Resuscitation Program.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for experienced providers include at least 3 years of pediatric and/or neonatal training, having previously performed >10 endotracheal intubations, and may include neonatologists, pediatric fellows, and neonatal nurse practitioners. Inclusion criteria for trainees: previous exposure to NRP, an interval of > 3 months elapsing between previous NRP applications, and may include pediatric residents, family medicine residents, nurses, respiratory therapists, neonatal fellows, and neonatal attendings.

Exclusion Criteria:

* Does not meet inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
No flow fraction | From start time of compression until 60 seconds have elapsed
  The proportion of time for which the mannequin received no effective compression (the number of seconds without effective chest compressions divided by the total number of seconds)

SECONDARY OUTCOMES:
Temperature regulation | From baseline to 30 seconds
  Infant placed in polyethylene wrap with warming mattress and hat placed on head.
Time of first heart rate check (seconds) | From baseline until heart rate check up to 5 minutes
  The number of seconds elapsed at the time the heart rate was first checked either by stethoscope, palpation of umbilical stump, or by EKG lead.
Heart rate check compliance | From baseline to 60 seconds up to 5 minutes
  HR was checked within 60 seconds after birth.
Time of bag mask ventilation (seconds) | From baseline to bag mask placement up to 5 minutes
  The number of seconds elapsed at the time the mask was first applied to the infant's face.
Bag mask ventilation compliance | From baseline to 60 seconds
  Mask was applied to the infant's face at 60 seconds after birth.
Time of sat probe placement (seconds) | From baseline to probe placement up to 5 minutes
  The number of seconds elapsed at the time the oxygen saturation probe was placed.
Sat probe placement compliance | From baseline to 60 seconds
  Sat probe placed at 60 seconds after birth.
Time of increase in FiO2 (seconds) | From simulation start to time of FiO2 increase up to 5 minutes
  The number of seconds elapsed at the time the amount of oxygen administered was increased.
MR SOPA Performance: Mask adjustment | From start of bag mask ventilation to 2 minutes
  Mask was adjusted on the infant's face
MR SOPA Performance: Reposition airway | From start of bag mask ventilation to 2 minutes
  infant's neck was adjusted
MR SOPA Performance: Suction mouth | From start of bag mask ventilation to 2 minutes
  infant's mouth was suctioned
MR SOPA Performance: Open mouth | From start of bag mask ventilation to 2 minutes
  infant's mouth was opened
MR SOPA Performance: Increased pressure | From start of bag mask ventilation to 2 minutes
  pressure on bag mask was increased
MR SOPA Performance: Placed advanced airway | From start of bag mask ventilation to 2 minutes
  endotracheal tube was placed
MR SOPA performed in correct sequence | From start of bag mask ventilation to 2 minutes
  corrective measures were performed in this sequence
MR SOPA measures all performed | From start of bag mask ventilation to 2 minutes
  each corrective measure was performed
Number of steps correctly performed | From start of bag mask ventilation to 2 minutes
  The number of steps correctly performed during the resuscitation
Time to effective ventilation (seconds) | From time of bag mask placement until chest rise up to 5 minutes
  The number of seconds elapsed at the time the mannequin had visible chest rise
Time to first compression (seconds) | From baseline until first compression up to 5 minutes
  The number of seconds elapsed at the time the first chest compression was performed
Correct hand position | From baseline until first compression up to 5 minutes
  Hands positioned with either two fingers on the mannequin's sternum or thumbs over the sternum with hands encircling the chest
Compression depth compliance | From baseline until first compression up to 5 minutes
  Compressions given at 1/3 of the infant's chest depth
Compression synchronization compliance | From start time of compression until 60 seconds have elapsed
  Synchronization with bag mask ventilation with a rate of 3 compressions: 1 ventilation
Compression rate per minute | From start time of compression until 10 seconds have elapsed
  Number of compressions within 10 seconds multiplied by 6
No blow fraction | From baseline to 10 minutes
  The proportion of time for which the mannequin received no effective ventilation (the number of seconds without effective ventilation divided by the total number of seconds)
Time to effective ventilation (seconds) | From baseline to time of first ventilated breath with an endotracheal tube up to 10 minutes
  The number of seconds elapsed at the time the mannequin is intubated and ventilated

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Gentle, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No